CLINICAL TRIAL: NCT06067113
Title: Hemodynamic and Functional Characteristics of the Cerebral Circulation in Obesity
Acronym: HemOB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Other Study IDs: PIC044-23_HRJC
Record Dates: First submitted 2023-08-18; First posted 2023-10-04 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-06

CONDITIONS: Cerebral Arterial Diseases
Keywords: Brain arteries; Brain hemodynamics; Obesity; Flow velocity; Vasoreactivity
MeSH Terms: conditions — Cerebral Arterial Diseases; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese: Obese patients with an indication for bariatric surgery
  Interventions: Procedure: Supraaortic and transcranial duplex
- Controls: Age and sex-matched controls
  Interventions: Procedure: Supraaortic and transcranial duplex

INTERVENTIONS:
Procedure: Supraaortic and transcranial duplex — Ecographic evaluation of supraaortic and transcranial arteries, including presence of plaques, flow velocities and pulsatility index
  Other Names: Brachial-ankle index; Brachial artery endothelium-dependent vasodilation

SUMMARY:
This prospective study is intended to explore differences in the cerebral hemodynamics and vascular functional characteristics between obese and normo-constituted patients; as well as the changes in the hemodynamic and functional characteristics in those same obese patients following the intense weight-loss that happens after bariatric surgery.

DETAILED DESCRIPTION:
Obesity, defined by the World Health Organization (WHO) as a body mass index of 30 or higher, is reaching epidemic proportions worldwide, with some 2.8 million attributable deaths annually. Initially linked to countries with higher incomes, it is now a serious health problem in countries with medium and low incomes.

The increase in body mass index from overweight to obesity is linearly correlated with an increase in coronary and cerebral vascular events, as well as death from vascular causes. Apart from the fact that obese patients are at higher risk of having classic vascular risk factors (independently associated with atherosclerosis and a risk of vascular events), the evident linear relationship between obesity and vascular pathology suggests the existence of pathophysiological mechanisms related to the accumulation of fat that cause structural and functional damage to the vascular system.

Adipokines are a group of pro-inflammatory peptides specifically secreted by fat tissue that have been linked to inflammatory activity, endothelial dysfunction, and insulin resistance in overweight and obese conditions. From these studies, a wealth of knowledge is drawn on the relationship of obesity with large-vessel atherosclerosis; but yet, few studies have focused on the particular relationship of obesity on the cerebral vasculature, despite the strong epidemiological relationship between obesity in middle age (and vascular risk factors in general) and cognitive deficits and vascular dementia in the elderly, possibly driven to a large extent by cerebral small vessel disease.

Small vessel disease (including both radiological signs on MRI in the form of white matter lesions, lacunar infarcts and/or cognitive impairment, and vascular dementia/Alzheimer's disease) have been positively correlated in several retrospective and prospective studies with the Gosling index or pulsatility index (PI) obtained by transcranial Doppler study in the middle cerebral artery. In recent years, much importance has been attached to the potential deleterious impact that small cerebral vessel disease in middle ages may have on degenerative brain diseases over 60 years of age, however, we have not identified a specific study of haemodynamic factors of cerebral circulation in middle-aged patients.

Obese patients with an indication for bariatric surgery constituted, in our opinion, an excellent model for the study of these potential haemodynamic factors (surrogate markers of subclinical cerebrovascular disease) in two ways: by comparing them with normal-constituted volunteers; as well as comparing them with themselves once they achieve an effective reduction in their body weight after surgery.

PRIMARY OBJECTIVE

To compare hemodynamic parameters of the cerebral circulation (mean arterial velocity and pulsatility index in the middle cerebral artery) of a sample of obese patients elective for bariatric surgery, in two ways: 1) with a sample of matched normal-weight volunteers by sex and age; 2) with themselves once they have achieved a loss of at least 25% of their original weight after surgery.

SECONDARY OBJECTIVES

To compare the following hemodynamic and functional indices between obese patients and normal-constituted volunteers, as well as between obese patients before and after losing at least 25% of their original weight after surgery:

DESCRIPTION OF THE INTERVENTION:

1. BASELINE VISIT

   The first visit (baseline visit) is similar for both patients and normal weight volunteers. It is divided into three parts:

   FIRST: interview with the patient to collect epidemiological and anthropometric data, including age, sex, height, weight, BMI, classic vascular risk factors, abdominal perimeter and drugs being taken.

   SECOND: the patient is instructed to lie down on the stretcher in a quiet environment with soft light in the room. After about 5 minutes of rest, blood pressure will be taken in the arms and legs for the subsequent calculation of the ankle-brachial index. Next, the endothelium-dependent vasodilation protocol will be carried out as follows: 1) initial measurement of the longitudinal diameter of the maximum brachial artery in systole from a frozen duplex image, in the middle third of one of the two arms (indistinctly); 2) a blood pressure cuff is placed on the same arm, which is inflated above 200 mm Hg (ensuring with a stethoscope that there is no tapping of the arterial pulse, or in other words, that effective ischemia occurs ). 3) Ischemia is maintained for 4 minutes using a stopwatch. 4) When the 4 minutes are up, the cuff is deflated and an attempt is immediately made to re-locate the brachial artery in a longitudinal section during the first minute releasing off the cuff; 5) one minute after deflating the cuff, with the artery already located, a measurement of the maximum diameter of the brachial artery in systole is taken again from a frozen image.

   THIRD PART: this last part consists of 4 parts:

   (A) Ultrasound study of supra-aortic trunks: IMT, mean arterial velocity and IP in terminal ACC and first segment of the cervical ICA after bifurcation.

   (B) Cannulation of a peripheral venous line. (C) Reconstitution of SONOVUE® contrast and administration of half the ampoule (the second half ampoule will be administered only in case all the desired measurements cannot be performed.

   (D) Transcranial duplex study with contrast, adjusting the power to acquire the following serial measurements:

   D.1 Peak-systolic, diastolic and mean arterial velocity in terminal ICA, middle segment of MCA, PCA-P1, ACA-A1 through transtemporal window of the most favorable side. Pulsatility index in the same arterial segments

   D2. Peak-systolic, diastolic and mean arterial velocity in the middle third of the basilar artery (BA) through transforaminal window. Pulsatility index in this segment.
2. FOLLOW-UP VISIT (PATIENTS ONLY)

   FIRST: interview with the patient to collect: weight, BMI, classic vascular risk factors, abdominal perimeter and drugs being taken.

   SECOND: the patient is instructed to lie down on the stretcher in a quiet environment with little light in the room. After a rest of about 5 minutes, blood pressure will be taken in the arms and legs for the subsequent calculation of the ankle-brachial index. Next, the endothelium-dependent vasodilation protocol will be carried out as follows: 1) initial measurement of the longitudinal diameter of the maximum brachial artery in systole from a frozen duplex image, in the middle third of one of the two arms ( indistinctly); 2) a blood pressure cuff is placed on the same arm, which is inflated above 200 mm Hg (ensuring with a stethoscope that there is no tapping of the arterial pulse, or in other words, that effective ischemia occurs ). 3) Ischemia is maintained for 4 minutes using a stopwatch. 4) When the 4 minutes are up, the cuff is deflated and an attempt is immediately made to re-locate the brachial artery in a longitudinal section during the first minute after deflating the cuff; 5) one minute after deflating the cuff, with the artery already located, a measurement of the maximum diameter of the brachial artery in systole is taken again from a frozen image.

   THIRD PART: this last part consists of 3 parts:

   (A) Ultrasound study of supra-aortic trunks: IMT, mean arterial velocity and IP in terminal ACC and first segment of the cervical ICA after bifurcation.

   (B) Cannulation of a peripheral venous line. (C) Reconstitution of the SONOVUE® contrast and administration of half the ampoule (the second half ampoule will be administered only in case all the desired measurements cannot be performed.

   (D) Transcranial duplex study with contrast, adjusting the power to acquire the following serial measurements:

   D.1 Peak-systolic, diastolic and mean arterial velocity in terminal ICA (ICA-T), middle segment of MCA, PCA-P1, ACA-A1 through transtemporal window of the most favorable side. Pulsatility index in the same arterial segments.

   D2. Peak-systolic, diastolic and mean arterial velocity in the middle third of the basilar artery (BA) through transforaminal window. Pulsatility index in this segment.

   DEVELOPMENT OF THE STUDY AND EVALUATION OF THE RESPONSE

   Recruitment will be carried out from the general surgery consultation, when it is decided to include the patient on the surgical waiting list, once the previous evaluation study has been completed and their suitability has been confirmed. At that time the possibility of participating in the study is explained to them. If the patient is interested, the general surgeon informs one of the study neurologists of this interest, who will contact him/her by telephone to offer further explanations about the type of study and possible discomfort caused orally, in addition to sending the informed consent via email. so you can read it calmly. If the patient decides to participate, she will communicate via email in response to the neurologist's initial sending with the signed and scanned informed consent, which will be saved in electronic format.

   Next, a day/time is agreed with the patient to carry out the initial visit. On that day, the patient will provide the signed informed consent in paper format, which will also be kept.

   Taking into account the sex and age characteristics of each of the patients, volunteers matched by age and sex with BMI below 25 will be recruited, recruited from the general neurology clinic or from non-blood relatives of the recruited patients. . In number of at least 10. The procedure and the tests to be performed will be the same as in the case of patients.

   GENERAL SCHEME

   VISIT 0 Patient Selection in General Cx consultations. Permission for telephone contact.

   VISIT 1 Telephone call to explain the study process and sending of informed consent by email, which must be signed and scanned and brought in person

   VISIT 2 Baseline Visit:
   * Clinical interview
   * Functional indices
   * Ultrasound study

   VISIT 3 Follow-up visit (applicable only to patients, at least 12 months after surgery and if they have lost at least 25% compared to initial weight):
   * Clinical interview
   * Functional indices
   * Ultrasound study

   EVALUATION OF RESULTS

   Primary Analysis

   Comparison of epidemiological variables, VAM, PI and functional indices (ankle-brachial index and endothelium-dependent vasodilation) between the group of obese patients before surgery and a group of normal weight volunteers, matched by sex and age. This will be done through a statistical analysis in three steps:
   * Descriptive analysis of both populations using measures of central tendency (proportions or standard deviations)
   * Univariate analysis using non-parametric tests
   * Logistic regression where the factors most related to obese patients or those clinically relevant are included, even if they do not meet the defined statistical criterion.

   Secondary analyzes

   Comparison of epidemiological variables, VAM, PI and functional indices between the group of obese patients before surgery and the same group at least 12 months after surgery and once they have lost at least 25% of their original weight. This will be done through a statistical analysis in three steps:
   * Descriptive analysis of both populations using measures of central tendency (proportions or standard deviations)
   * Univariate analysis using non-parametric tests
   * Logistic regression where the factors most related to obese patients or those clinically relevant are included, even if they do not meet the defined statistical criterion.

   ADVERSE EVENTS

   This is an observational study without active intervention. The only potential risks are described below and are not considered slight or minor in all cases:
   * The derivatives of the canalization of a peripheral venous access can be pain and hemorrhages, in both cases located in the puncture area and temporary.
   * The risks derived from the administration of eco-enhancers are mild and temporary. Nausea, vomiting, headaches, altered taste, dizziness and skin rashes have been reported. Serious adverse reactions such as hypotension, bronchospasm and urticaria have been described in 0.001-0.006% of patients.
   * The risks associated with performing the endothelium-dependent vasodilation study due to controlled ischemia in one arm are local pain and ecchymosis, both temporary.

   No adverse effects have been described after performing cervical or transcranial ultrasound.

   ETHICAL ASPECTS

   GENERAL AND SPECIFIC RULES FOR RESEARCHERS

   The researchers will strictly adhere to the provisions of this protocol, properly completing the data collection notebooks. The study will be carried out in accordance with the recommendations contained in the Declaration of Helsinki, revised at successive world assemblies (last in Fortaleza, Brazil, October 2013) and the Standards of Good Clinical Practice.

   The research team (recruitment, explanation and procedures with patients, anonymization) is made up of members of the General Surgery and Endocrinology and Nutrition services, in addition to Dr. Álvaro Bonelli Franco of Neurology. The data analyzes will be performed blindly by Drs. Teresa Montalvo and Jose Fdez. Ferro from the Neurology service.

   INFORMED CONSENT All patients will be informed before starting the study of the objectives and procedures that will be carried out. The patient information sheet and informed consent models appear in Annex 1 and 2 of this protocol.

   SECURITY AND CONFIDENTIALITY DEVICES The information disseminated and obtained by the implementation of this study is considered confidential and will be treated at all times in accordance with Organic Law 3/2018, of December 5, on the Protection of Personal Data and guarantee of digital rights and in Regulation (EU) 2016/679 of the European Parliament and of the Council of 04/27/2016. An Excel database will be created specifically designed for the study, in which patients will be identified with a numerical code assigned in order of recruitment, and which will not contain personal information about the patients.

   SURE The only interventions that the patient will be subjected to during the study are venipuncture, the infusion of potentiators and the performance of a transient ischemia in one arm, all of them considered very low-cost interventions, therefore, they are not considered It is necessary to take out civil liability insurance.

   ECONOMIC MEMORY

   This study arises from an independent initiative of the researchers. No type of financial remuneration is contemplated either for the patient or for the study researchers. To cover the expenses derived from the use of eco-enhancers (Sonovue®) as well as the costs of writing and translating the manuscript for a potential competitive publication of the results, the project will be submitted to research aid competitions where appropriate.

   PRACTICAL CONSIDERATIONS

   Researchers will adhere to the standards of Good Clinical Practice. All information collected during the study will be recorded directly in the attached data collection notebook. When a correction is made, the date and initials of the person making it must be noted. Prior to the study, the patient must receive oral and written information regarding the design, purposes of the study and possible risks that may arise from it. If they subsequently agree to participate in it, they must sign their consent, without this preventing them from revoking it at any time and for any reason and abandoning the study. Patients will be instructed regarding the need to strictly follow the investigators' instructions. Patients will be informed of the need to contact the researchers if any incident arises during the study, providing them with how to do so.

   There will be an electronic documentation file for all data, which will be kept intact for ten years after completion of the study.

   STATISTIC ANALYSIS

   SAMPLE SIZE The absence of previous studies makes it difficult to calculate the sample size following a rigorous statistical method. We have thought about including 15 patients with obesity, estimating a 20% loss during follow-up for various reasons (revocation of their participation during follow-up or not achieving the minimum weight loss estimated a priori despite the surgery, which we set in 25%). We believe that the differences between patients and healthy controls, as well as between patients before and after losing weight, will be considerable in both hemodynamic and functional factors to observe differences with this number of participants, in view of the published observational studies. previously.

   STATISTIC ANALYSIS It will be carried out with the appropriate statistical techniques for the prespecified study variables. A descriptive analysis of the population is carried out. Frequency results will be expressed in absolute terms, as percentages and confidence intervals. Continuous variables will be expressed as mean (SD) and median (range) according to the normality test (Kolmogorov Smirnov test). To study the relationship between the different variables, Chi square or Analysis of Variance will be used if they are parametric. And if a normal distribution is not followed, a non-parametric test will be used (Mann-Whitney U or Kruskal Wallis, as appropriate). The SPSS 18 statistical package (SPSS Inc. Chicago, IL, USA) will be used.

ELIGIBILITY:
INCLUSION CRITERIA

* Morbid obesity (BMI above 40) or a BMI of 35 and obesity-related health conditions
* Indication for bariatric surgery as losing weight treatment
* Sign informed consent

EXCLUSION CRITERIA

* Age under 18 years or over 59 years
* Pregnancy
* Patients with acute heart disease
* Denial or withdrawal of the informed consent
* Absence of acoustic window despite the use of eco-enhancers.
* Inability to channel a peripheral line.
* The subject fails to achieve, after surgery, a weight loss of at least 25% of the initial weight

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients between 18 and 59 years with morbid obesity and an indication for bariatric surgery after evaluation by the hospital's interdisciplinary commission, who are included on the surgical waiting list.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean flow velocity in middle cerebral artery | through study completion, an average of 1 year
  Mean flow velocity in middle cerebral artery

SECONDARY OUTCOMES:
Ankle-brachial index | through study completion, an average of 1 year
  Index calculated with arterial pressure measurements in the arm, knee and ankle
Intima-media thickness in distal CCA | through study completion, an average of 1 year
  Intima-media measures in the distal common carotid artery
Endothelium-dependent brachial artery vasodilation | through study completion, an average of 1 year
  Rate of change in the brachial after a 4 minute complete occlusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Rey Juan Carlos, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
This is specifically specified in the informed consent to patients.

REFERENCES:
- [Background] Frosen J, Joutel A. Smooth muscle cells of intracranial vessels: from development to disease. Cardiovasc Res. 2018 Mar 15;114(4):501-512. doi: 10.1093/cvr/cvy002. PMID 29351598
- [Result] Hubert HB, Feinleib M, McNamara PM, Castelli WP. Obesity as an independent risk factor for cardiovascular disease: a 26-year follow-up of participants in the Framingham Heart Study. Circulation. 1983 May;67(5):968-77. doi: 10.1161/01.cir.67.5.968. PMID 6219830
- [Result] Fantuzzi G, Mazzone T. Adipose tissue and atherosclerosis: exploring the connection. Arterioscler Thromb Vasc Biol. 2007 May;27(5):996-1003. doi: 10.1161/ATVBAHA.106.131755. Epub 2007 Feb 15. PMID 17303782
- [Result] Kidwell CS, el-Saden S, Livshits Z, Martin NA, Glenn TC, Saver JL. Transcranial Doppler pulsatility indices as a measure of diffuse small-vessel disease. J Neuroimaging. 2001 Jul;11(3):229-35. doi: 10.1111/j.1552-6569.2001.tb00039.x. PMID 11462287
- [Result] Ghorbani A, Ahmadi MJ, Shemshaki H. The value of transcranial Doppler derived pulsatility index for diagnosing cerebral small-vessel disease. Adv Biomed Res. 2015 Feb 17;4:54. doi: 10.4103/2277-9175.151574. eCollection 2015. PMID 25802823
- [Result] Mok V, Ding D, Fu J, Xiong Y, Chu WW, Wang D, Abrigo JM, Yang J, Wong A, Zhao Q, Guo Q, Hong Z, Wong KS. Transcranial Doppler ultrasound for screening cerebral small vessel disease: a community study. Stroke. 2012 Oct;43(10):2791-3. doi: 10.1161/STROKEAHA.112.665711. Epub 2012 Sep 4. PMID 22949475
- [Result] Foerstl H, Biedert S, Hewer W. Multiinfarct and Alzheimer-type dementia investigated by transcranial Doppler sonography. Biol Psychiatry. 1989 Oct;26(6):590-4. doi: 10.1016/0006-3223(89)90084-x. PMID 2790097
- [Result] Harris S, Reyhan T, Ramli Y, Prihartono J, Kurniawan M. Middle Cerebral Artery Pulsatility Index as Predictor of Cognitive Impairment in Hypertensive Patients. Front Neurol. 2018 Jul 20;9:538. doi: 10.3389/fneur.2018.00538. eCollection 2018. PMID 30083126
- See also: WHO | 10 facts on obesity. — http://www.who.int/news-room/facts-in-pictures/detail/6-facts-on-obesity